CLINICAL TRIAL: NCT06261918
Title: Transcriptional and Epimetabolic Profile of Breast Carcinoma With Luminal or HER2+ or Locally Advanced Triple-negative Histotype in Patients With/Without Previous Clinical History of Metabolic Syndrome
Acronym: PROMETA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FABI ALESSANDRA, Prof.ssa, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6269
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Metabolic Syndrome
MeSH Terms: conditions — Breast Neoplasms; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without metabolic syndrome: Pre/postmenopausal patients diagnosed with breast cancer undergoing NCT and subsequent surgery with long follow-up
  Interventions: Procedure: Influence of metabolic syndrome on the achievement of pathological complete response
- Patients with metabolic syndrome: Pre/postmenopausal patients diagnosed with breast cancer undergoing NCT and subsequent surgery with long follow-up
  Metabolic syndrome evaluated on the basis of the following criteria:
  1. BMI≥30
  2. Glycosylated hemoglobin/baseline blood glucose
  3. Triglycerides
  4. Hypertension
  5. Lipid profile
  Interventions: Procedure: Influence of metabolic syndrome on the achievement of pathological complete response

INTERVENTIONS:
Procedure: Influence of metabolic syndrome on the achievement of pathological complete response — The proposed activity aims to assess the transcriptional and epimetabolic profile of locally advanced luminal or HER2+ or triple negative breast cancer in patients with/without metabolic syndrome to predict the therapeutic response to neoadjuvant chemotherapy.

SUMMARY:
This prospective pilot study of biological specimens aims to identify new prognostic and predictive biomarkers of response to standard therapy for local advanced BC, as well as to identify new targets for the development of immuno- therapeutic protocols. First aim is therefore to expand our knowledge to increase the response to preoperative treatment, intensify treatment patterns, and select patients based on clinical parameters. In this regard, it appears imperative to investigate yet under-investigated factors that might impair the response to standard therapy for local advanced BC including association to metabolic syndrome and analysis of tumoral and stromal features supporting a tumor microenvironment impenetrable to both drugs and immune system cells.

DETAILED DESCRIPTION:
Breast cancer (BC) represents the most common cancer disease among women. In Italy, according to the Aiom-Airtum Report "Cancer Numbers 2020," there are an estimated 54,976 new cases in the female population, which represents 30.3 % of all cancers. Although adherence to screening programs has improved in recent years, the diagnosis of locally advanced BC accounts for about 30% of new diagnoses.

Neo-adjuvant therapy (NCT), which is the administration of chemotherapy drugs combined with biologic therapies if indicated, is the gold-standard in the setting of patients with locally advanced BC (1). It allows down-staging of the primary neoplasm so that conservative rather than demolitive surgical treatment can be performed. NCT also allows prognostic evaluation based on the response obtained to the treatment itself. Noteworthy, a large meta-analysis conducted on 11955 patients enrolled in 12 different clinical trials reported a significant correlation between obtaining a pathological complete response (pathological complete response, pCR, i.e., absence of invasive disease in both breast and lymph nodes) and both event-free survival (EFS) and overall survival (OS) in all tumor subtypes, albeit more pronounced for HER-2 positive neoplasms (EFS: HR 0. 39, CI 95% 0.31-0.50; OS: HR 0.34, CI 95% 0.24-0.47) or triple negative (EFS: HR 0.24, CI 95% 0.18-0.33; OS: HR 0.16, CI 95% 0.11-0.25) (2). To date, about 30% of BC patients go on to pCR following NCT (2), thus highlighting the need for further investigation to expand the proportion of these patients who may benefit from long-lasting clinical responses following such therapy. The consideration of a preexisting history of metabolic syndrome might open new avenues in therapeutic and prognostic perspectives.

Despite the numerous drugs currently available for the NCT, classic chemotherapy (CT) represents the most widely used class of drugs. Growing pieces of evidence show that the efficacy of CT depends not only on its ability to directly inhibit or kill malignant cells, but also on features of the tumor microenvironment in term of metabolic alterations, which might influence the anti-tumoral response (3). Specifically, tumor cell death promoted by cytotoxic drugs causes the release of cancer-associated antigens that, in turn, activate and recruit immune cells within the tumor (4). A recent Italian phase 2 study, the GIADA trial, showed that the number of tumor-infiltrating lymphocytes is significantly associated with pCR and that anthracycline-based chemotherapy treatment results in the establishment of a more immunogenic tumor microenvironment (5). Early results show that despite an improvement in pCR, a considerable number of treated individuals still do not respond or lack long-term responses (6). This evidence suggests that such combinatorial regimens often fail to neutralize all of the immunosuppressive activities that BC enacts to resist CT, evade the anti-tumor immune response, and progress (7). To date, the identification of a system that can predict responses to NCT and the delineation of mechanisms of immunosuppressive resistance in patients with BC unresponsive to NCT remain unresolved issues.

The complex network of interactions between immune cells and other components of the tumor microenvironment results in significant heterogeneity in clinical practice to the response to precision medicine therapeutic options. Consequently, it will be increasingly important to decipher the functional status of the metabolic status of the tumor microenvironment in each patient in order to move from standardized therapy to individualized treatment that in the future could increase survival and improve the quality of life of a greater numbers of BC patients.

ELIGIBILITY:
Inclusion Criteria:

Patients will be treated as per standard. Inclusion criteria depend exclusively on compliance with informed consent, tumor size (only advanced stage tumors will be used for the study) and histological diagnosis. Specifically, patients with the following will be included in the proposed study:

* Histological diagnosis of locally advanced Luminal or HER2+ or Triple negative breast cancer (cT2, T3, T4 N0 or any T N1, N2, N3, M0), clinical stage II to III disease.
* Age > 18 years
* Regular clinical and instrumental follow up
* Informed consent form signed by enrolled patients - Availability of information from medical records:

  1. pre/post NAC blood chemistry tests: blood count, glycemia/glycosylated hemoglobin, lipid profile (triglycerides, total cholesterol, HDL + LDL cholesterol);
  2. BMI;
  3. possible therapy with oral hypoglycaemic drugs/insulin; statins; diuretics/antihypertensive drugs;
  4. Sex hormone hormonal status (pre- or post-menopause);

Exclusion Criteria:

* Prior or synchronous history of systemic malignancy. - History of homo- or contralateral breast cancer.
* Evidence of metastatic (Stage IV) disease.
* Neo-adjuvant treatment with hormonal therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre/postmenopausal patients diagnosed with breast cancer undergoing NCT and subsequent surgery with long follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Acheivement of pathological complete response | 36 months
  The presence of metabolic syndrome or lifestyle influences the achievement of the full pathological response

SECONDARY OUTCOMES:
Event-free survival (EFS) | 36 moths
  The presence of metabolic syndrome or lifestyle can reduce the development of cancer recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli - IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No